CLINICAL TRIAL: NCT02537535
Title: Guidelines Oriented Approach to Lipid Lowering (GOAL) in Canada
Acronym: GOAL
Status: Completed | Type: Observational
Sponsor: Canadian Heart Research Centre (Other)
Collaborators: Amgen (Industry)
Responsible Party: Principal Investigator, Dr. Anatoly Langer, Anatoly Langer, MD, M.Sc., FRCP (C), FACC -Chair, Canadian Heart Research Centre, Canadian Heart Research Centre
Other Study IDs: CHRC2014-GOAL Canada Study
Record Dates: First submitted 2015-08-26; First posted 2015-09-01 (Estimated); Last update posted 2020-01-23 (Actual); Status verified 2020-01

CONDITIONS: Dyslipidemia
MeSH Terms: conditions — Dyslipidemias | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: survey — This is a cross-sectional study without specific intervention

SUMMARY:
Cross-sectional observational study designed to identify and describe the care gap in guideline-oriented low density lipoprotein cholesterol (LDL-C) management in Canadian patients at high cardiovascular risk.

DETAILED DESCRIPTION:
This is a cross-sectional observational study designed to provide real-life data on the current management of dyslipidemia in high cardiovascular risk patients in routine clinical practice. Canadian guidelines recommend a target for LDL-C of ≤2.0 mmol/L (or ≥50% decrease) after treatment initiation in high-risk patients. The recommended first line treatment is statin therapy. Available data clearly indicates that up to 50% of high risk patients do not achieve this important target because of statin inadequacy or intolerance leading to non-adherence.

Therefore this program aims to provide further insights into the challenges Canadian physicians face in helping their high risk patients achieve guideline-recommended LDL-C.

ELIGIBILITY:
Inclusion Criteria:

1. Adults ≥ 18 years old 2. High risk for cardiovascular morbidity and mortality (at least one of the following):

1. Clinical vascular disease:

   * Coronary Artery Disease (CAD): history of myocardial infarction (MI), Coronary artery bypass grafting (CABG), percutaneous coronary intervention (PCI), angiographic disease
   * Cerebrovascular Disease (CeVD): history of cerebrovascular accident (CVA) or transient ischemic attack (TIA), carotid surgery
   * Abdominal Aortic Aneurism (AAA): history of surgery/intervention
   * Peripheral Arterial Disease (PAD): history of surgery/intervention
2. Familial hypercholesterolemia defined as LDL-C > 5 mmol/L and one of:

   * typical physical findings (stigmata) such as tendon xanthomata, xanthelasma, and arcus corneae
   * personal history of early cardiovascular disease
   * family history of early cardiovascular disease or of marked hyperlipidemia
3. Receiving current optimal (maximal or maximal tolerated) statin therapy for at least 3 months prior to patient enrolment
4. LDL-C > 2.0 mmol/L measured within 6 months of patient enrolment date and while on (despite) maximal tolerated statin therapy (± other lipid modifying therapies).
5. Desire and ability to execute the consent to participate.

Exclusion criteria:

1. Current treatment with PCSK9 inhibitor
2. Participation in an investigational study
3. Prior participation in the GOAL program

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Low density lipoprotein cholesterol (LDL-C) management in Canadian patients at high cardiovascular risk
Sampling Method: Non-Probability Sample
Enrollment: 2027 (Actual)
Dates: Start 2016-01 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Mean LDL-C level according to lipid lowering treatment received | up to 2 years
  defined as: a. Prior cardiovascular disease, b. "High risk" Diabetes (as per Canadian Diabetes Association Guidelines), c. High risk patients based on Framingham score; and according to LDL-C between 2.5 and 3.0 mmol/L and LDL > 3.0 mmol/L

SECONDARY OUTCOMES:
Mean LDL-C level in patients with Familial Hypercholesterolemia | up to 2 years
Mean LDL-C level in patients with statin intolerance | up to 2 years
Mean LDL-C level in patients receiving combination dyslipidemia therapy | up to 2 years
Mean LDL-C level according to statin efficacy | up to 2 years
  according to patient's statin efficacy (high, moderate, etc. by dose)
Mean LDL-C level according to their type of medication insurance coverage | up to 2 years

IPD SHARING:
Plan to Share IPD: No